CLINICAL TRIAL: NCT01817244
Title: A Long Term Effect of Collaborative Care on Depression Treatment in a Community Dwelling Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Clinical Research Coordination Center, Seoul, Korea (Other Government)
Responsible Party: Principal Investigator, Hyeon Woo Yim, Professor, National Clinical Research Coordination Center, Seoul, Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A102065_2013
Record Dates: First submitted 2013-03-13; First posted 2013-03-25 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Depression
Keywords: care management; depression; elderly; Korea
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- care management type 1 (Experimental): 2-month care management
  Interventions: Other: care management
- care management type 2 (Active Comparator): 6-month care management
  Interventions: Other: care management

INTERVENTIONS:
Other: care management — 6-month care management

SUMMARY:
Suicide is a significant cause of death in Korea. According to the report compiled by the Korea National Statistical Office, 24.8 victims of every 100,000 in 2007 (Korea National Statistical Office, 2008), which is higher compared with 10.1 in the United States, 6.0 in the United Kingdom, and 19.1 in Japan (Organisation for Economic Co-operation and Development, 2008). Especially, suicide rate is incredibly higher in elderly. Most persons who commit suicide have a diagnosed psychiatric disorder. Among them, 60% had Depression when they committed suicide. Therefore, this study aimed the impact of a care management intervention on depression treatment and reducing suicidal ideation in elderly patients with depression.

ELIGIBILITY:
Inclusion Criteria:

* 60 and older
* current major or minor depression

Exclusion Criteria:

* severe cognitive dysfunction
* severe auditory dysfunction
* history of psychosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAMD) | 6 months after baseline

SECONDARY OUTCOMES:
suicide ideation | 6 months after baseline
  suicide ideation: suicide questionnaire
treatment compliance | at 6 months from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Kunkuk University of Chungju Hospital, Chungju, Choong-Book, South Korea